CLINICAL TRIAL: NCT01337310
Title: A Phase I Study of Tesetaxel Administered Once Every 21 Days to Japanese Subjects With Advanced Solid Tumors
Brief Title: Study of Tesetaxel in Japanese Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOPK106
Record Dates: First submitted 2011-04-04; First posted 2011-04-18 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced solid tumors
MeSH Terms: interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tesetaxel (Experimental): Tesetaxel administered orally once every 21 days for at least 2 cycles
  Interventions: Drug: Tesetaxel

INTERVENTIONS:
Drug: Tesetaxel — The starting dose for the first 3 patients treated will be 24 mg/m2. In the absence of dose-limiting toxicity, the dose will be increased by 3 mg/m2 for the next group of 3 patients treated. Interpatient dose escalation will continue in this manner to 27 and 31 mg/m2 until the maximum tolerated dose or the maximum dose allowed per protocol (31 mg/m2) is reached and 6 patients are treated at this dose.
  Other Names: DJ-927

SUMMARY:
Tesetaxel is an orally active tubulin-binding inhibitor of the taxane class. Evaluation of tesetaxel in Japanese patients has been limited. This study is being conducted to determine the maximum tolerated dose and safety of tesetaxel administered orally once every 21 days to Japanese patients.

ELIGIBILITY:
Primary inclusion criteria:

* At least 20 years of age
* Morphologic or cytologic confirmation of an advanced or metastatic solid tumor malignancy, not to include lymphoma, for which no standard therapy exists or for which resistance or intolerance to standard therapy has developed
* ECOG performance status not more than 1
* Adequate bone marrow, hepatic, and renal function
* Willing to remain hospitalized for at least 10 days following tesetaxel administration in Cycle 1
* At least 4 weeks and recovery from effects of prior surgery or other therapy with an approved or investigational agent, with resolution of any toxicity to not more than Grade 1

Primary exclusion criteria:

* Brain metastasis or leptomeningeal disease
* Significant medical disease other than cancer
* Neuropathy greater than Grade 1

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose in mg/m2 based on the dose-limiting adverse events that occur | First cycle (expected to be 21 days, including the day of first dose of tesetaxel followed by a rest period)

SECONDARY OUTCOMES:
Dose-limiting toxicities (adverse events that result in a reduction in the dose of tesetaxel in the dose-escalation scheme) | First cycle (expected to be 21 days, including the day of first dose of tesetaxel followed by a rest period)
Percentage of patients with adverse events | Through 30 days after the last dose of tesetaxel
Tumor response rate | After Cycle 2 (expected to be after Day 42 counting from the date of first dose of tesetaxel)

CONTACTS AND LOCATIONS:
Locations (1):
- Kinki University School of Medicine, Osaka-fu, Japan